CLINICAL TRIAL: NCT04104100
Title: Prevalence and Risk Factors of Nocturnal Polyuria in Women With Lower Urinary Tracts Symptoms Based on Bladder Diary
Brief Title: Prevalence and Risk Factor of NP in Women With LUTS
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907002RIN
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-08

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Nocturnal polyuria; Bladder diary
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with nocturnal polyuria: Nocturnal polyuria was defined when the proportion of night-time voided volume over 24-hour voided volume was greater than 33% for ≥65 year-old women, and when the proportion of night-time voided volume over 24-hour voided volume was greater than 20% for <65 year-old women.
- Women without nocturnal polyuria: Nocturnal polyuria was defined when the proportion of night-time voided volume over 24-hour voided volume was greater than 33% for ≥65 year-old women, and when the proportion of night-time voided volume over 24-hour voided volume was greater than 20% for <65 year-old women.

SUMMARY:
The knowledge of prevalence and risk factors of nocturnal polyuria might be important for the treatment of women with lower urinary tract symptoms (LUTS). Thus, our aim is to describe the prevalence and risk factors of nocturnal polyuria in women with LUTS.

DETAILED DESCRIPTION:
Between September 2010 and January 2019, all women with LUTS visiting urogynecological department of a medical center for urodynamic evaluation were reviewed. Nocturnal polyuria was defined when the proportion of night-time voided volume over 24-hour voided volume was greater than 33% for ≥65 year-old women, and when the proportion of night-time voided volume over 24-hour voided volume was greater than 20% for <65 year-old women. Backward stepwise multivariable logistic regression analysis was performed using all statistical variables in the univariate logistic regression analysis. P < 0.05 was considered as statistical significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with lower urinary tract symptoms
* Complete a 3-day bladder diary

Exclusion Criteria:

* <20 y/o or > 85 y/o
* Regular urethral catheterization or intermittent self-catheterization
* Urinary tract infection or chronic inflammation in the previous 2 weeks
* Bladder calculus
* Neurogenic bladder due to radical hysterectomy or injury of the central nervous system
* History of pelvic radiotherapy or a preexisting malignant pelvic tumor.

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with lower urinary tract symptoms
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Nocturnal polyuria | Between August 2007 and December 2010
  Nocturnal polyuria was defined when the proportion of night-time voided volume over 24-hour voided volume was greater than 33% for ≥65 year-old women, and when the proportion of night-time voided volume over 24-hour voided volume was greater than 20% for <65 year-old women.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, PhD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Hashim H, Blanker MH, Drake MJ, Djurhuus JC, Meijlink J, Morris V, Petros P, Wen JG, Wein A. International Continence Society (ICS) report on the terminology for nocturia and nocturnal lower urinary tract function. Neurourol Urodyn. 2019 Feb;38(2):499-508. doi: 10.1002/nau.23917. Epub 2019 Jan 15. PMID 30644584
- [Background] Hofmeester I, Kollen BJ, Steffens MG, Bosch JL, Drake MJ, Weiss JP, Blanker MH. Impact of the International Continence Society (ICS) report on the standardisation of terminology in nocturia on the quality of reports on nocturia and nocturnal polyuria: a systematic review. BJU Int. 2015 Apr;115(4):520-36. doi: 10.1111/bju.12753. Epub 2015 Jan 26. PMID 24684483